CLINICAL TRIAL: NCT02623985
Title: Evaluation of Accuracy of Rapid Tests for Group A Beta Hemolytic Streptococci in Out-patients With Sore Throat From Acute Pharyngitis at Siriraj Hospital
Brief Title: Evaluation of Accuracy of Rapid Tests for Group A Beta Hemolytic Streptococci in Out-patients With Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Adhiratha Boonyasiri, Dr., Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 539-2558-EC1
Record Dates: First submitted 2015-11-26; First posted 2015-12-08 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sofia (Experimental): Patients who presented with sore throat will be performed throat swab and sent for Sofia which is rapid test.
  Interventions: Device: Sofia
- QuickVue (Experimental): Patients who presented with sore throat will be performed throat swab and sent for QuickVue which is rapid test.
  Interventions: Device: QuickVue
- Throat swab culture (Experimental): Patients who presented with sore throat will be performed throat swab and sent for throat swab culture which is gold standard.
  Interventions: Device: Throat swab culture

INTERVENTIONS:
Device: Sofia — Patients who presented with sore throat will be performed throat swab and sent for Sofia for rapid test.
  Other Names: Sofia for rapid test
  Arms: Sofia
Device: QuickVue — Patients who presented with sore throat will be performed throat swab and sent for QuickVue for rapid test.
  Other Names: QuickVue for rapid test
  Arms: QuickVue
Device: Throat swab culture — Patients who presented with sore throat will be performed throat swab and sent for throat swab culture for gold standard.
  Other Names: throat swab culture for gold standard
  Arms: Throat swab culture

SUMMARY:
The purpose of this study is to evaluate accuracy of rapid tests for group A beta hemolytic streptococci in patients who presented with sore throat at out patient department in Siriraj Hospital.

DETAILED DESCRIPTION:
The patients who presented with sore throat at out patient department less than 5 days and age over 6 years old would be enrolled by the primary physicians and the consent forms will be completed by researcher.

The throat swab would be performed by using Sofia, QuickVue rapid tests compare to the gold standard which is a throat swab culture to evaluate the accuracy of the rapid tests.

The sample size for validation of sensitivity and specificity of rapid tests is 358 patients.

The primary outcome is will be evaluated sensitivity and specificity of both rapid tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients who came with sore throat less than 5 days.

Exclusion Criteria:

* No

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Of participants positive for Group A Streptococcus by Sofia rapid test, the percentage who are positive for Group A Streptococcus by Sofia rapid test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 95% confidence limits.
Of participants positive for Group A Streptococcus by Sofia rapid test, the percentage who are negative for Group A Streptococcus by Sofia rapid test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 95% confidence limits.
Of participants positive for Group A Streptococcus by QuickVue rapid test, the percentage who are positive for Group A Streptococcus by QuickVue rapid test. | Day 1
  Establish sensitivity against a gold standard. Report as a percentage of participants with 95% confidence limits.
Of participants positive for Group A Streptococcus by QuickVue rapid test, the percentage who are negative for Group A Streptococcus by QuickVue rapid test. | Day 1
  Establish specificity against a gold standard. Report as a percentage of participants with 95% confidence limits.

REFERENCES:
- [Background] Plainvert C, Duquesne I, Touak G, Dmytruk N, Poyart C. In vitro evaluation and comparison of 5 rapid antigen detection tests for the diagnosis of beta-hemolytic group A streptococcal pharyngitis. Diagn Microbiol Infect Dis. 2015 Oct;83(2):105-11. doi: 10.1016/j.diagmicrobio.2015.06.012. Epub 2015 Jun 23. PMID 26159722